CLINICAL TRIAL: NCT06623617
Title: A Study on the Three-Dimensional Breathing Patterns of Patients With Postpartum Stress Urinary Incontinence Based on Pelvic Diaphragm Dynamics
Brief Title: Three-Dimensional Breathing Patterns in Postpartum Stress Urinary Incontinence
Acronym: PPSUI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jie Li (Other)
Responsible Party: Sponsor-Investigator, Jie Li, Nurse, Shenzhen Hospital of Southern Medical University
Organization: Shenzhen Hospital of Southern Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JieLi
Record Dates: First submitted 2024-09-28; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: Three-Dimensional Breathing; Postpartum Stress Urinary Incontinence; elvic Diaphragm Dynamics; pelvic floor exercises
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group：three-dimensional breathing training group (Other): Engage in app-based three-dimensional breathing training and learn to use a biofeedback pressure device at home for proper and effective training. They will also be guided to log their daily training, manually inputting data such as duration and frequency. A virtual assistant will provide real-time feedback based on this data, including encouragement and adjustments to training intensity.
  Interventions: Behavioral: Three-dimensional breathing training; Behavioral: control group：Health education
- Control group：Health education (Other): The control group received health education, which was conducted one-on-one by researchers during the recruitment of mothers. The content included the etiology and risk factors of PPSUI (Prolapse of Pelvic Organs during Straining), the benefits and precautions of pelvic floor muscle exercises and breathing, as well as the implementation methods.
  Interventions: Behavioral: control group：Health education

INTERVENTIONS:
Behavioral: Three-dimensional breathing training — Engage in app-based three-dimensional breathing training and learn to use a biofeedback pressure device at home for proper and effective training. They will also be guided to log their daily training, manually inputting data such as duration and frequency. A virtual assistant will provide real-time feedback based on this data, including encouragement and adjustments to training intensity.
  Arms: Intervention Group：three-dimensional breathing training group
Behavioral: control group：Health education — Provide participants with health education, which is conducted one-on-one by researchers during the recruitment of mothers. The content includes the etiology and risk factors of PPSUI (Pelvic Organ Prolapse during Straining), the benefits and precautions of pelvic floor muscle exercises and breathing techniques, as well as the implementation methods.

SUMMARY:
**Clinical Trial** The purpose of this clinical trial is to determine whether three-dimensional breathing training is effective in treating postpartum stress urinary incontinence (PPSUI). The main question it aims to answer is: Can three-dimensional breathing training improve or treat postpartum stress urinary incontinence?

Participants will:

* Receive one-on-one verbal health education covering the causes and risk factors of PPSUI, benefits and precautions of pelvic floor exercises and breathing, and implementation methods.
* Engage in app-based three-dimensional breathing training and learn to use a biofeedback pressure device at home for proper and effective training. They will also be guided to log their daily training, manually inputting data such as duration and frequency. A virtual assistant will provide real-time feedback based on this data, including encouragement and adjustments to training intensity.

DETAILED DESCRIPTION:
User Experience Quality Control

1. Establish a dedicated technical team for system testing and quality control to ensure stable operation of the APP and accurate data.
2. Regularly update and optimize the virtual characters to guarantee the best user experience.

Data Security and Privacy Protection

1. Ensure that all user data is encrypted to protect user privacy and data security.
2. Comply with relevant regulations and standards to ensure the lawful use and protection of user data.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 20-35 years
2. Postpartum: 42 to 49 days
3. Diagnosed with pure postpartum stress urinary incontinence (PPSUI) by an experienced obstetrician/gynecologist during the first postpartum check-up, according to the International Continence Society (ICS) standards.

Exclusion Criteria:

1. BMI > 30 kg/m²
2. Cesarean section
3. Multiparous women
4. Pathological conditions or deformities of the spine
5. History of lumbopelvic surgery
6. Urogenital prolapse of grade 2 or higher
7. Professional athletes
8. Severe cardiopulmonary conditions during pregnancy or postpartum
9. Neurological diseases or cognitive impairments
10. Individuals unable to meet study requirements

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Rate of Treatment for PPSUI Patients | The measurement is conducted 8 weeks after the intervention.
  Criteria for Cure: Both no leakage on the ICIQ-SF assessment and a negative Stress Induced Test must be met.
  Criteria for Improvement: A reduction of ≥1 point in the frequency dimension score or a reduction of ≥2 points in the volume dimension score on the ICIQ-SF assessment after treatment.
  Criteria for Ineffectiveness: No change or an increase in the scores of both the frequency and volume dimensions of urine leakage on the ICIQ-SF assessment.

SECONDARY OUTCOMES:
Pelvic Floor Muscle Strength | The measurement is conducted 8 weeks after the intervention.
  Pelvic Floor Muscle Strength: Assessed using the modified Oxford grading system.
  0 level (no muscle activity),
  1. level (only muscle tremors or pulsations),
  2. level (muscle strength can be felt but there is no lifting or squeezing sensation),
  3. level (muscle strength is greater than level 2, lifting sensation can be felt; at this point, muscle contraction can be observed visually, and when 3 levels or above are detected, the examiner presses the posterior vaginal wall with their finger to provide resistance),
  4. level (muscle strength is increased and contractions are good, capable of lifting the posterior vaginal wall against resistance),
  5. level (capable of lifting the posterior vaginal wall against resistance, with the therapist's index and middle fingers being pinched together and pinched together and pulled towards the vagina).
Pelvic Floor Ultrasound Assessment of the Anterior Compartment | The measurement is conducted 8 weeks after the intervention.
  he ultrasonic diagnostic criterion for cystocele is when the lowest point of the bladder reaches the level of or below the reference line during maximum Valsalva maneuver. Further distinction of cystocele subtypes is made according to the Green classification criteria: Type I: Posterior vesicourethral angle ≥ 140°, urethral rotation angle < 45°; Type II: Posterior vesicourethral angle ≥ 140°, urethral rotation angle ≥ 45°; Type III: Posterior vesicourethral angle < 140°, urethral rotation angle ≥ 45°.
Degree of Anterior and Middle Compartment Prolapse | The measurement is conducted 8 weeks after the intervention.
  Using the Pelvic Organ Prolapse Quantification (POP-Q) system, the degree of pelvic prolapse is assessed by measuring the distances between indicator points on the anterior wall, posterior wall, and apex of the vagina [two points on the anterior wall (Aa, Ba), two points on the posterior wall (Ap, Bp), and two points on the apex (C, D)] and the hymenal plane. Additionally, the genital hiatus, perineal body, and vaginal length are recorded to reflect the pelvic prolapse condition. In this study, we focused on the anterior compartment values that are more relevant to PPSUI (Pelvic Organ Prolapse Surgical Site Infection). Measurements were taken at the initial visit and at the end of treatment. Specifically, patients were positioned in the lithotomy position and instructed to perform a Valsalva maneuver to measure anterior vaginal wall prolapse (if a Valsalva maneuver could not be elicited at the initial visit, the assessment was conducted after initial treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Wenzhi First Name: （Wenzhi） Middle initial: （） Degree: （Professor）, Study Chair — Shenzhen Hospital of Southern Medical University

IPD SHARING:
Plan to Share IPD: No